CLINICAL TRIAL: NCT04771065
Title: Microendoscopic Transventricular Deep Brain Stimulation of the Anterior Nucleus of the Thalamus as a Safe and Efficient Treatment in Intractable Epilepsy
Brief Title: Deep Brain Stimulation of the Anterior Nucleus of the Thalamus in Intractable Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0106
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Refractory Epilepsy
Keywords: epilepsy; deep brain stimulation; thalamus; endoscopy; stereotaxy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Deep Brain Stimulation (DBS) of the anterior nucleus of the thalamus (ANT) has been proposed in patients with severe intractable epilepsy. When used, the transventricular approach increases the risk of bleeding due the anatomy around the entry point in the thalamus. To avoid such a complication, the investigators used a transventricular microendoscopic technique.

ELIGIBILITY:
Inclusion criteria:

* adult patients
* treated between 2010 and 2019 for refractory epilepsy by DBS of the anterior nucleus os the thalamus using microendoscopy
* minimum follow-up of 1-year
* refractory epilepsy defined as failure of at least 3 antiepileptic drugs

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients extracted from our prospective database, who have been surgically treated between 2010 and 2019 for refractory epilepsy by deep brain stimulation (DBS) of the anterior thalamic nucleus using microendoscopy. All patients had a minimum follow up of 1 year. Refractory epilepsy was defined as failure of at least 3 anti-epileptic drugs (AEDs) to produce adequate seizure control
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Absence of hemorraghic complication | 1 day
  Absence of hemorraghic complication on post operative MRI

SECONDARY OUTCOMES:
responder rate | 1 year
  50%-responder rate (on seizures)
responder rate | 2 years
  50%-responder rate (on seizures)
responder rate | 5 years
  50%-responder rate (on seizures)

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Poulen, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC